CLINICAL TRIAL: NCT00679614
Title: The Effect of the Combined Use of Naloxone and Tramacet on Postoperative Analgesia in Elderly Patients Having Joint Replacement Surgery: a Randomized Controlled Study.
Brief Title: Effect of Combined Use of Naloxone and Tramacet on Postop Analgesia in Elderly Patients Having Joint Replacement Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-07-427; 13659
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Hip Arthroplasty; Knee Arthroplasty; Spinal Anesthesia
Keywords: Tramacet; naloxone; morphine; analgesia; elderly; elderly patients
MeSH Terms: conditions — Agnosia | interventions — Naloxone; Ultracet; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Group A oral tramacet 2 tablets preoperatively, 2 tablets every 6 hours for 5 days then 1-2 tablets of tramacet prn to a maximum of 8 tablets per day. Naloxone infusion starting preop at 0.25ug/kg/hr and continuing during hospital stay (an equivalent of 400ug over 24 hours in a 70 kg man). The infusion will be discontinued 1 hour before patient discharge.
  Interventions: Drug: tramacet, naloxone
- 2 (Active Comparator): Group B will receive oral tramacet 2 tablets preoperatively and then 2 tablets every 6 hours for five days. ( or until discharge. Patient VAS after discontinuation of morphine PCA may dictate addition of oral narcotic oxycodone after discharge). This group will also receive saline infusion at 4-6mls / hour for the duration of the hospital stay.
  Interventions: Drug: tramacet
- 3 (Active Comparator): Group C will receive oral Acetaminophen tablets 1 gm preoperatively and subsequently 6 hourly plus an infusion of saline (placebo) at a rate of 4-6mls / hour for the duration of their stay.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: tramacet, naloxone — Group A: oral tramacet 2 tablets preoperatively, then 2 tablets every 6 hours for 5 days then 1-2 tablets of tramacet prn to a maximum of 8 tablets per day. A naloxone infusion will started preop at 0.25ug/kg/hr and will continue during patient's stay in hospital (an equivalent of 400ug over 24 hours in a 70 kg man). Infusion discontinued 1 hour before patient discharge. All the patients in groups A and B will be provided Morphine PCA for the duration of their hospital stay. Use of morphine PCA will be noted.Oral celebrex 200mg will be given to all the patient twice a day for five days as per our standard practice. All patients will receive peri-articular infiltration with local anesthetic solution intraoperatively by the surgeon as per our standard practice.
  Other Names: tramadol/acetaminophen
  Arms: 1
Drug: tramacet — Group B: oral tramacet 2 tablets preop,then 2 tablets every 6 hours for five days(or until discharge. Patient VAS after discontinuation of morphine PCA may dictate addition of oral narcotic oxycodone after discharge). Group also receives saline infusion at 4-6mls/hour during hospital stay.All patients in groups A and B will have Morphine PCA during hospital stay. Use of morphine PCA will be noted. Oral celebrex 200mg will be given to all the patient twice a day for five days as per our standard practice. All patients will receive peri-articular infiltration with local anesthetic solution intraopby the surgeon as per our standard practice.
  Other Names: tramadol/acetaminophen
  Arms: 2
Drug: Acetaminophen — Group C will receive oral Acetaminophen tablets 1 gm preoperatively and subsequently 6 hourly plus an infusion of saline (placebo) at a rate of 4-6mls / hour for the duration of their stay. Oral celebrex 200mg will be given to all the patient twice a day for five days as per our standard practice. All patients will receive peri-articular infiltration with local anesthetic solution intraoperatively by the surgeon as per our standard practice. The Visual Analogue Scale, the Ramsay Sedation Score and the Mini Mental State Exam will be used to assess the patients for pain, sedation and confusion every 6 hours while in hospital.
  Other Names: Tylenol
  Arms: 3

SUMMARY:
Patients over 70 years of age, scheduled for joint replacement surgery will be randomized to tramacet/ naloxone plus morphine PCA or to morphine PCA to assess quality of analgesia in the postoperative period.

The primary objective is to determine opioid use during combined use of oral tramacet and naloxone infusion perioperatively in elderly patients (70 yrs and older) having elective knee/ hip arthroplasty under spinal anesthesia.

Secondary objectives are to determine the incidence VAS scores ≥4 and adverse effects such as nausea, vomiting, sedation, respiratory depression, pruritus, confusion, and time of independent mobilization.

Hypothesis: Perioperative naloxone infusion and tramacet provides adequate analgesia in elderly patients undergoing total knee/hip arthroplasty and is associated with 80% reduction in opioid use and reduced opioid-induced side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 70 years and older*
2. Able to give informed consent
3. Able to communicate in English
4. Having elective hip/knee arthroplasty
5. ASA physical status 1-3.

Exclusion Criteria:

1. Allergies to any of the following: naloxone, tramacet, NSAIDs, or local anesthetic
2. Contraindication to spinal anesthesia
3. Contraindication to use of tramacet or celebrex
4. ASA physical status 4
5. Chronic opioid use
6. Chronic pain syndrome All the above will be included in the letter of information

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-12-17 (Actual); Primary Completion 2011-05-31 (Actual); Study Completion 2011-05-31 (Actual)

PRIMARY OUTCOMES:
Morphine use / day | per day

CONTACTS AND LOCATIONS:
Overall Officials: Ngozi Imasogie, MBBS, FRCA UK, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- St Joseph's Health Care, London, Ontario, Canada